CLINICAL TRIAL: NCT06589323
Title: Cardiac Surgery Residents' Learning Curve of Intraoperative Transit-time Flowmetry and High-frequency Ultrasound in Coronary Artery Bypass Surgery: the LEARNERS Study
Brief Title: Residents' Learning Curve of Intraoperative Transit-time Flowmetry and High-frequency Ultrasound in CABG (LEARNERS)
Acronym: LEARNERS
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Federico Cammertoni, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6735
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: adult patients undergoing coronary artery bypass surgery
  Interventions: Procedure: Coronary artery bypass graft

INTERVENTIONS:
Procedure: Coronary artery bypass graft — All patients included will undergo coronary artery bypass graft surgery. During surgery, every graft will be evaluated through transit time flowmetry (TTFM) and intraoperative ultrasound control (HFUS).

SUMMARY:
Transit-time flowmetry (TTFM) allows grafts quality assessment during coronary artery bypass surgery by measuring the flow volume through them. Recently the intraoperative epicardial high-frequency ultrasound (HFUS) was introduced, with the possibility of capturing bidimensional images of the anastomoses. When combined, these two techniques provide high diagnostic yield reaching a positive predictive value of 100 percent.

Despite current guidelines recommend the employment of TTFM and HFUS, they remain largely underused probably because of limited information and the lack of standardization. Furthermore, surgeons must overcome a learning curve to handle both techniques properly, but few data are available according the current literature.

The main purpose of this study is to evaluate the complexity of HFUS and TTFM learning curve. This is a prospective, observational, monocentric cohort study. Adult patients undergoing coronary artery bypass surgery will be enrolled.

DETAILED DESCRIPTION:
This is a prospective, observational, monocentric cohort study in which adult patients undergoing coronary artery bypass surgery will be enrolled.

Primary objective of this study is to evaluate the complexity of cardiac surgery residents' learning curve for grafts quality assessment with transit-time flowmetry (TTFM) and intraoperative epicardial high-frequency ultrasound (HFUS).

Secondary objectives are to evaluate the complexity of cardiac surgery residents' learning curve for grafts quality assessment with TTFM and HFUS as isolated techniques.

The study will last four months (three months for patients enrollment and data collection and one month for statistical analysis and scientific paper writing).

The trial will start after obtaining favourable opinion from the local Ethics Committee and could be considered completed when all the eight cardiac surgery residents involved have reached primary endpoint.

All patients with coronary artery disease and an indication for surgical revascularization (coronary artery bypass grafting) who meet the above-described inclusion and exclusion criteria will be enrolled by signing the informed consent the day before surgery.

Patient data (anamnestic data, surgery description, intraoperative echographic and flowmetric measurements) will be recorded in a dedicated database. All data recorded in the database are commonly acquired for all patients undergoing this type of surgery and no further examinations will be performed for patients included in the trial.

The study will involve cardiac surgery residents with different levels of training and an expert cardiac surgeon who acts as supervisor and benchmark. Each resident will sign a dedicated informed consent form in the presence of a doctor foreign to the study protocol (Cardiac Surgery ward cardiologist). The residents will be "blinded" about the trial objective and the adopted score system. They will undergo a specific training including a quick lesson and a practical workshop to familiarize with the equipment.

During surgery, every graft will be evaluated through transit time flowmetry (TTFM) and intraoperative ultrasound control (HFUS).

In details, the ultrasound control is carried out through a dedicated sterile ultrasound probe connected to a machine (MiraQ - MEDISTIM) as soon as each anastomosis is completed. The result of the evaluation is recorded together with surgery data. This evaluation is intended to confirm the correct realization of the anastomosis and provides a proof of its patency.

Once each graft is completed, the resident will be given 60 seconds to acquire two HFUS recordings (short and long axis). After that, the supervisor will perform his personal recording which will stand as benchmark. The following items will be evaluated:

A) Long axis recording acquired within 60 seconds [YES-> 1] [NO -> 0] B) Long axis recording judged as suitable by the supervisor [YES -> 1] [NO -> 0] C) Short axis recording acquired within 60 seconds [YES -> 1] [NO -> 0] D) Short axis recording judged as suitable by the supervisor [YES -> 1] [NO -> 0]

E) Correct interpretation of the anastomosis as adequate or inadequate [YES -> no penalty] [NO -> total score becomes 0 and the resident isn't allowed to perform TTFM]

Each resident will be given a HFUS-related score from a minimum of 0 to a maximum of 4.

Whenever one of the recordings will be judged as non-suitable by the supervisor and consequently useless for a correct interpretation of the anastomosis (score 0 for items A and/or C), item E won't be evaluated and the HFUS will be given a total score of 0.

Next step will be the TFM evaluation, which is carried out through a specific sterile device connected to the same machine (MiraQ - MEDISTIM) once the patient has been weaned from the cardiopulmonary bypass and before protamine administration. This recording is performed under EKG and pressure-controlled conditions. Although there is no general agreement on the optimal mean arterial pressure at which the measurement has to be recorded, the investigators will adopt the standard used in the REQUEST study protocol (16), that is an average pressure of 80 mmHg.

The resident will acquire the TTFM recording after each graft is completed. To make the comparison as accurate as possible, the resident will perform TTFM evaluation on one graft at a time and successively the supervisor will do the same for each graft (making sure that delta between the pressure during the two recordings is lower than 10 percent and that no drug has been administered). The following items will be evaluated:

F) Time necessary to acquire the measures [< 30 sec -> 1] [> 30 sec, < 60 -> 0.5] [> 60 sec -> 0] G) Need for multiple measurements before the final one: [>2 -> 0] [1 -> 0.5] [ 0 -> 1] H) Need to change probe dimensions: [NO -> 0] [YES-> 1]

I) ACI [delta between resident and supervisor measurements < 10%-> 1] [> 10%, < 20% -> 0.5] [> 20% -> 0] L) Mean Flow [delta between resident and supervisor measurements < 10%-> 1] [> 10%, < 20% -> 0.5] [> 20% -> 0] M) Pulsatility Index [delta between resident and supervisor measurements < 10%-> 1] [> 10%, < 20% -> 0.5] [> 20% -> 0] N) Backward Flow [delta between resident and supervisor measurements < 10%-> 1] [> 10%, < 20% -> 0.5] [> 20% -> 0] O) Diastolic Filling [delta between resident and supervisor measurements < 10%-> 1] [> 10%, < 20% -> 0.5] [> 20% -> 0]

P) Correct interpretation of the graft quality as working [YES -> no penalty] [NO -> total score becomes 0]

Each resident will be given a TTFM-related score from a minimum of 0 to a maximum of 8.

The final score for each graft will be the sum of the two scores (HFUS and TTFM), from a minimum of 0 to a maximum of 12.

The same procedure will be repeated for each graft performed during the surgery.

Each resident will continue until reaching a ratio between total score and number of evaluated anastomoses of 11.

Our cardiac surgery unit performs between 5 and 10 coronary artery bypass grafts surgeries per week on average. Considering the inclusion and exclusion criteria and assuming that some patient may not give their informed consent, the investigators expect to enroll 4 patients per week. Considering that the involved residents (8 in total) will take part to the procedures in turn and that around 10 surgeries are needed to become autonomous, the investigators estimate to enroll 80 patients during a period of 3 months.

Data will be collected in a specific database (Microsoft Excel worksheet). The Kolgomorov-Smirnoff test was used to check for variables distribution. Continuous variables with a normal distribution are summarized by mean and standard deviation. Continuous variables with a non-normal distribution are expressed with median and interquartile range.

Categorical variables are reported as absolute frequency distribution and percentage. Continuous data are analyzed using the unpaired t-test or the Mann - Whitney test according to their distribution. Categorical data are compared with the Fisher's exact test. Statistical findings were considered significant if p value was less than 0.05. Statistical analysis will be performed with the statistic software SPSS (IBM).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old;
* Written informed consent;
* Indication to CABG surgery (both "on-pump" and "off-pump");
* Stable angina, unstable angina or acute coronary syndrome without ST elevation (NSTEMI).

Exclusion Criteria:

* Age >= 18 years old;
* Written informed consent;
* Indication to CABG surgery (both "on-pump" and "off-pump");
* Stable angina, unstable angina or acute coronary syndrome without ST elevation (NSTEMI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with coronary artery disease and an indication for surgical revascularization (coronary artery bypass grafting) who meet the above-described inclusion and exclusion criteria will be enrolled by signing the informed consent the day before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Number of anastomoses needed to reach a ratio (total score/n. of anastomoses) >= 11 | This evaluation will require from 1 to 3 months.
  Number of anastomoses needed to reach a ratio between total score and the number of studied anastomoses of 11 or more

SECONDARY OUTCOMES:
Number of anastomoses needed to reach a ratio (HFUS score/n. of anastomoses) = 4 | This evaluation will require from 1 to 3 months.
  Number of anastomoses needed to reach a ratio between the HFUS score and the number of studied anastomoses of 4
Number of anastomoses needed to reach a ratio (TTFM score/n. of anastomoses) >=7 | This evaluation will require from 1 to 3 months.
  Number of anastomoses needed to reach a ratio between the TTFM score and the number of studied anastomoses of 7 or more

CONTACTS AND LOCATIONS:
Overall Officials: Federico Cammertoni, Dr., Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Result] Kieser TM, Rose S, Kowalewski R, Belenkie I. Transit-time flow predicts outcomes in coronary artery bypass graft patients: a series of 1000 consecutive arterial grafts. Eur J Cardiothorac Surg. 2010 Aug;38(2):155-62. doi: 10.1016/j.ejcts.2010.01.026. Epub 2010 Feb 21. PMID 20176493
- [Result] Kieser TM, Taggart DP. The use of intraoperative graft assessment in guiding graft revision. Ann Cardiothorac Surg. 2018 Sep;7(5):652-662. doi: 10.21037/acs.2018.07.06. PMID 30505750
- [Result] Amin S, Pinho-Gomes AC, Taggart DP. Relationship of Intraoperative Transit Time Flowmetry Findings to Angiographic Graft Patency at Follow-Up. Ann Thorac Surg. 2016 May;101(5):1996-2006. doi: 10.1016/j.athoracsur.2015.10.101. Epub 2016 Feb 12. PMID 26876343
- [Result] Di Giammarco G, Pano M, Cirmeni S, Pelini P, Vitolla G, Di Mauro M. Predictive value of intraoperative transit-time flow measurement for short-term graft patency in coronary surgery. J Thorac Cardiovasc Surg. 2006 Sep;132(3):468-74. doi: 10.1016/j.jtcvs.2006.02.014. PMID 16935097
- [Result] Xenogiannis I, Zenati M, Bhatt DL, Rao SV, Rodes-Cabau J, Goldman S, Shunk KA, Mavromatis K, Banerjee S, Alaswad K, Nikolakopoulos I, Vemmou E, Karacsonyi J, Alexopoulos D, Burke MN, Bapat VN, Brilakis ES. Saphenous Vein Graft Failure: From Pathophysiology to Prevention and Treatment Strategies. Circulation. 2021 Aug 31;144(9):728-745. doi: 10.1161/CIRCULATIONAHA.120.052163. Epub 2021 Aug 30. PMID 34460327
- [Result] Di Giammarco G, Canosa C, Foschi M, Rabozzi R, Marinelli D, Masuyama S, Ibrahim BM, Ranalletta RA, Penco M, Di Mauro M. Intraoperative graft verification in coronary surgery: increased diagnostic accuracy adding high-resolution epicardial ultrasonography to transit-time flow measurement. Eur J Cardiothorac Surg. 2014 Mar;45(3):e41-5. doi: 10.1093/ejcts/ezt580. Epub 2013 Dec 12. PMID 24335472
- [Result] Gaudino M, Sandner S, Di Giammarco G, Di Franco A, Arai H, Asai T, Bakaeen F, Doenst T, Fremes SE, Glineur D, Kieser TM, Lawton JS, Lorusso R, Patel N, Puskas JD, Tatoulis J, Taggart DP, Vallely M, Ruel M. The Use of Intraoperative Transit Time Flow Measurement for Coronary Artery Bypass Surgery: Systematic Review of the Evidence and Expert Opinion Statements. Circulation. 2021 Oct 5;144(14):1160-1171. doi: 10.1161/CIRCULATIONAHA.121.054311. Epub 2021 Oct 4. PMID 34606302
- [Result] Kieser TM. Graft quality verification in coronary artery bypass graft surgery: how, when and why? Curr Opin Cardiol. 2017 Nov;32(6):722-736. doi: 10.1097/HCO.0000000000000452. PMID 28806185
- [Result] Andreasen JJ, Nohr D, Jorgensen AS, Haahr PE. Peroperative epicardial ultrasonography of distal coronary artery bypass graft anastomoses using a stabilizing device. A feasibility study. J Cardiothorac Surg. 2020 Jan 8;15(1):3. doi: 10.1186/s13019-020-1057-x. PMID 31915030
- [Result] Andreasen JJ, Nohr D, Jorgensen AS. A case report on epicardial ultrasonography of coronary anastomoses using a stabilizing device without the use of ultrasound gel. J Cardiothorac Surg. 2019 Mar 13;14(1):59. doi: 10.1186/s13019-019-0882-2. PMID 30866994
- [Result] Wolf RK, Falk V. Intraoperative assessment of coronary artery bypass grafts. J Thorac Cardiovasc Surg. 2003 Sep;126(3):634-7. doi: 10.1016/s0022-5223(03)00747-5. No abstract available. PMID 14502132
- [Result] Budde RP, Meijer R, Dessing TC, Borst C, Grundeman PF. Detection of construction errors in ex vivo coronary artery anastomoses by 13-MHz epicardial ultrasonography. J Thorac Cardiovasc Surg. 2005 May;129(5):1078-83. doi: 10.1016/j.jtcvs.2004.09.002. PMID 15867783
- [Result] Jorgensen AS, Schmidt SE, Staalsen NH, Ostergaard LR. An Improved Algorithm for Coronary Bypass Anastomosis Segmentation in Epicardial Ultrasound Sequences. Ultrasound Med Biol. 2016 Dec;42(12):3010-3021. doi: 10.1016/j.ultrasmedbio.2016.07.014. Epub 2016 Sep 2. PMID 27592558
- [Result] Taggart DP, Thuijs DJFM, Di Giammarco G, Puskas JD, Wendt D, Trachiotis GD, Kieser TM, Kappetein AP, Head SJ. Intraoperative transit-time flow measurement and high-frequency ultrasound assessment in coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2020 Apr;159(4):1283-1292.e2. doi: 10.1016/j.jtcvs.2019.05.087. Epub 2019 Aug 22. PMID 31685277
- [Derived] Cammertoni F, Di Giammarco G, Testa N, Pavone N, Marcolini A, D'Avino S, Bruno P, Grandinetti M, Bianchini F, Trapani AE, Massetti M. Learning Curve of Cardiac Surgery Residents in Transit-Time Flow Measurement and High-Resolution Epicardial Ultrasonography During Coronary Surgery. J Clin Med. 2026 Jan 13;15(2):620. doi: 10.3390/jcm15020620. PMID 41598558

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT06589323/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT06589323/ICF_001.pdf